CLINICAL TRIAL: NCT04888338
Title: Outcomes After Chimeric Antigen Receptor Therapy (CAR-T) and Radiation Therapy (RT) for Hematologic Malignancies
Brief Title: Outcomes After Chimeric Antigen Receptor Therapy and Radiation Therapy for Hematologic Malignancies
Status: Recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-1150; NCI-2021-00910 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2020-1150 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2021-02-24; First posted 2021-05-17 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Hematopoietic and Lymphoid Cell Neoplasm
MeSH Terms: conditions — Hematologic Neoplasms | interventions — Electronic Health Records

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational (data collection): Patients medical records are reviewed for details about CAR-T and RT treatment and acute and late toxicities, disease outcomes such as any events related to local or distant disease progression, survival, and cause of death if available. Patients' imaging scan data is collected at baseline, within 2 months of the first treatment of RT or CAR-T, and at 3, 6, 12 months, and then annually for 5 years after RT completion.
  Interventions: Other: Data Capture; Other: Electronic Medical Record

INTERVENTIONS:
Other: Data Capture — Treatment related data is collected
Other: Electronic Medical Record — Medical records are reviewed
  Other Names: Computer Based Patient Record; EMR; EMR (electronic medical record)

SUMMARY:
This study collects information on outcomes after chimeric antigen receptor therapy and radiation therapy for hematologic malignancies. Collecting information from patients before, during, and after receiving chimeric antigen receptor therapy or radiation therapy may help doctors to optimize patient selection, dose, timing, and sequencing of these treatments.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Record clinical outcomes of patients with hematologic malignancies receiving standard-of-care chimeric antigen receptor therapy (CAR-T) nd/or standard-of- care bispecific therapy, and radiation therapy (RT).

SECONDARY OBJECTIVES:

I. To record patient-specific factors and treatment-related factors in patients with hematologic malignancies receiving standard-of-care CAR-T, and/or standard-of-care bispecific therapy, and RT to ultimately improve patient selection and overall treatment strategy to optimize clinical outcomes. II. To record and explore the relationship between radiation dose, target, technique, and timing with respect to CAR-T, and/or standard-of-care bispecific therapy and clinical outcomes in patients with hematologic malignancies treated with standard-of-care CAR-T, and/ or standard-of-care bispecific therapy, and RT.

III. To record and study the relationship between patient-specific factors and treatment-related factors and treatment toxicity in patients with hematologic malignancies undergoing standard-of-care CAR-T, and/or standard-of-care bispecific therapy, and RT.

OUTLINE:

Patients medical records are reviewed for details about CAR-T and RT treatment and acute and late toxicities, disease outcomes such as any events related to local or distant disease progression, survival, and cause of death if available. Patients' imaging scan data is collected at baseline, within 2 months of the first treatment of RT or CAR-T, and at 3, 6, 12 months, and then annually for 5 years after RT completion.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Treatment with or intention to treat with radiation therapy, standard-of-care CAR-T cell therapy and/or standard-of-care bispecific therapy, within a 90 day window for a hematologic malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are receiving CAR-T cell therapy or radiation therapy for hematologic malignancy
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-04-10 (Actual); Primary Completion 2026-11-14 (Estimated); Study Completion 2026-11-14 (Estimated)

PRIMARY OUTCOMES:
Clinical outcomes of patients with hematologic malignancies receiving standard-of-care chimeric antigen receptor therapy (CAR-T) and radiation therapy (RT) | Up to 5 years
  Outcome measures will include the following: date and type of disease progression, time to lymphoma progression, progression confirmed on biopsy (yes/no), disease control within the radiation field, survival and date of death, cause of death, overall response rate/best response achieved, duration of response, Toxicities including adverse events (CTCAE v 5.0), Neurotoxicity (ICANS) and cytokine release syndrome grade

SECONDARY OUTCOMES:
Patient-specific factors and treatment-related factors | Up to 5 years
  Patient- and treatment-related outcome measures include the following: Type of hematologic malignancy, disease stage, presence of bulky and/or extranodal disease, number of prior lines of therapy, treatment with prior stem cell transplant, radiation treatment dose/fractionation, target, technique, timing of radiation relative to CAR-T cell therapy, type of CAR-T cell therapy, bridging and conditioning therapy received, laboratory studies including LDH and CRP
Relationship between radiation dose, target, technique, and timing with respect to CAR-T and clinical outcomes | Up to 5 years
  "Correlation between radiation dose, target, technique, and timing with respect to CAR-T and clinical outcomes." Radiation details include the following: radiation treatment dose/fractionation, target, technique, timing of radiation relative to CAR-T cell therapy, radiation treatment intent. Clinical outcome measures include the following: date and type of disease progression, time to lymphoma progression, progression confirmed on biopsy (yes/no), disease control within the radiation field, survival and date of death, cause of death, overall response rate/best response achieved, duration of response, Toxicities including adverse events (CTCAE v 5.0), Neurotoxicity (ICANS) and cytokine release syndrome grade
Relationship between patient-specific factors and treatment-related factors and treatment toxicity | Up to 5 years
  Patient and treatment-related factors include the following: Type of hematologic malignancy, disease stage, presence of bulky and/or extranodal disease, number of prior lines of therapy, treatment with prior stem cell transplant, radiation treatment dose/fractionation, target, technique, timing of radiation relative to CAR-T cell therapy, type of CAR-T cell therapy, bridging and conditioning therapy received, laboratory studies including LDH and CRP Treatment toxicity includes the following: adverse events (CTCAE v 5.0), Neurotoxicity (ICANS) and cytokine release syndrome grade

CONTACTS AND LOCATIONS:
Overall Officials: Penny Q Fang, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center website — http://www.mdanderson.org